CLINICAL TRIAL: NCT00064545
Title: Gene-by-Smoking Interactions and Risk of Atherosclerosis - Ancillary to ARIC
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kari North, PhD, Associate Professor, University of North Carolina, Chapel Hill
Other Study IDs: 1227; 5R01HL074377 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-10 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Carotid Artery Diseases; Peripheral Vascular Diseases; Cerebral Arteriosclerosis; Cerebrovascular Accident
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Carotid Artery Diseases; Peripheral Vascular Diseases; Intracranial Arteriosclerosis; Stroke

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate common genetic variations, that in combination with exposure to tobacco smoke, may modify the risk of atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

While cigarette smoking is a well-established and potent risk factor for atherosclerotic vascular disease, individual susceptibility to smoking varies considerably, suggesting modifiers such as genomic variation. Several key enzymes involved in the activation and detoxification of mutagenic tobacco smoke compounds, oxidative stress, and DNA damage are expressed in the tissues of the heart and vasculature and represent mechanistic pathways for tobacco-induced pathology. Many of these enzymes have common polymorphisms (greater than or equal too 10% prevalence in the population) with known functional effects. Although restricted to a few enzymes and hampered by shortcomings in design, a small number of studies have suggested that enzymatic activation and detoxification of tobacco smoke modifies the risk of certain cardiovascular outcomes associated with cigarette smoking.

DESIGN NARRATIVE:

The genetic epidemiology study will evaluate common genetic polymorphisms that, in combination with exposure to tobacco smoke, may modify the risk of atherosclerosis and its clinical sequelae. An average of six polymorphisms, selected on the basis of their prevalence and functional significance, expression in relevant tissues, evaluation in previous studies and biologic plausibility, within 19 genes involved in activation, detoxification, oxidative stress, and DNA repair pathways will be evaluated as an ancillary study to the Atherosclerosis Risk in Communities (ARIC) study. In this well-characterized, bi-ethnic cohort of 15,792 men and women under active follow-up since 1987-89 (completeness of follow-up 96%), five endpoints quantifying subclinical atherosclerosis and validated clinical atherosclerotic events will be studied in case-cohort/case-control mode: incident coronary heart disease, carotid atherosclerosis, peripheral arterial disease, incident stroke, and MRI-detected cerebral infarcts. The study is well designed to study how DNA sequence polymorphisms can promote or inhibit the atherogenic effects of smoking and the risk of clinical events, and to contribute new knowledge on the role of genetic variation in the response to environmental insults and toxicants.

A case-cohort or case-control approach will be taken, using data from the Atherosclerosis Risk in Communities (ARIC) study. Approximately 20 polymorphisms will be examined in relation to five cardiovascular disease (CVD) endpoints. The polymorphisms to be examined are classified as variants of either a) Phase I (activation) enzymes, b) Phase II (detoxification) enzymes, c) oxidative stress enzymes, or d) DNA repair enzymes. The CVD endpoints include incident coronary heart disease (CHD) cases (n=1,101), incident stroke cases (n=323), prevalent peripheral artery disease (PAD) (n=237 cases), carotid atherosclerosis determined by MRI (n=504 cases), and cerebral infarcts (n=237cases). Controls will consist of 1,062 controls selected at visit 1, and 237 visit-3 controls for the cerebral infarct cases. The statistical approach will be based on the proportional hazards regression for incident CHD and stroke endpoints, and logistic regression for the other CVD outcomes. Both additive and multiplicative forms of interaction will be tested.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ARIC cohort, incident cases of CHD and cohort representative sample.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
CHD | Baseline - 2001

CONTACTS AND LOCATIONS:
Overall Officials: Kari North, Principal Investigator — University of North Carolina, Chapel Hill